CLINICAL TRIAL: NCT00956501
Title: Assessment of Postural Orientation and Equilibrium In Early Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 02-09-12B
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2013-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: fall; balance
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this pilot study is to characterize changes in postural orientation and equilibrium in early diagnosed ALS patient. The investigators plan to cross validate the use of a standardized test of equilibrium (EquiTest, Computerized Dynamic Posturography - CDP) in early diagnosed ALS patients.

DETAILED DESCRIPTION:
ALS is a progressive neurodegenerative disorder involving primarily upper and lower motor neurons. The progressive loss in motor neurons leads to weakness, fatigue, spasticity, and loss of balance. Falls are reported in 30-35% of ALS patients prior to enrolment to ALS clinic. This early loss of balance may not be detected by the classical neurological exam, or the standard clinical balance scales. Understanding the impairments in the balance control system which leads to fall during the course of ALS is a prerequisite for the clinical decision-making process in order to develop a proper balance rehabilitation program and fall prevention strategies for these patients.

Patients and control subjects will undergo balance system evaluation consisting of the following testing:

1. Sensory Organization Test Protocol

   Standardized EquiTest assessment protocol:

   Sensory Organization Test (SOT) - will be used to measure change how well participants maintain balance under progressively more difficult test conditions, which either disrupt or remove visual and proprioceptive feedback. Visual and proprioceptive environments will be altered systematically for fixed support and sway-referenced support and surround conditions, and under normal (eyes open), absent (eyes closed), and sway-referenced vision (eyes sway-referenced). Under sway-referenced conditions, the platform on which the subject stands and/or the visual surround also move proportionally to their AP sway. During SRC the floor and visual surround are controlled by a servomechanism (Gain=1.0) to follow movements of the subjects' center of gravity. Sway-referencing eliminates accurate somatosensory and/or visual information used to orient the body. Performance under sway-referenced visual conditions shows the participant's ability to suppress conflicting visual inputs and to rely on alternative systems for maintaining equilibrium (table 1).

   Participants are carefully positioned on the platform by aligning the lateral malleoli with the axis of rotation of the platform and visual surround. Participants wear a harness during all testing, which protects participants from falling. As an additional safety measure, the technician stands behind the participant. There are three trials per condition with each trial lasting 20 seconds. When a participant takes a step, touches the surround panels, or needs assistance from the technician, that trial is marked as a fall and the participant receives an equilibrium score of zero for that trial.

   In addition to the ES, movement strategy scores (MSS) will be measured by horizontal shear forces. Movement strategy scores reflect the relative use of movement about the ankle, hips and upper body to maintain balance during the SOT. Scores around 100 reflect a predominant use of ankle strategy to maintain balance, whereas low scores are indicative of the use of hip strategies to restore stability.
2. Motor Control Test Protocol The Motor Control Test (MCT), using the same apparatus will be performed to examine postural responses to external perturbations. During the MCT, subjects will receive perturbation from the force platform. Perturbations are expressed as translation movement (medium horizontal anterior to posterior movements of less than 1 sec. duration) or as rotation movements (at 6.0 degrees per second, which cause ankle dorsiflexion or plantarflexion). Six forward and six backward translations are generated. Five toes up and five toes down rotations are generated. The computer assures random delays of 1.5 to 2.5 seconds between translation trials and 3.0 to 5.0 seconds between rotation trials. During each perturbation, the computer monitors the subjects sway responses, measuring forces exerted against the dual force plate. These forces are expressed as weight symmetry and strength symmetry. Weight symmetry measures the distribution of total body weight over each leg, independent of other response strength and strength symmetry measures. Weight symmetry scores near 100 indicate a symmetrical weight distribution (EquiTest manual, 1991).

Outcome variables:

i. Sensory Organization Test (SOT) scores on conditions 1-6. ii. Movement Strategy Score on conditions 1-6 iii. Weight Symmetry Score on conditions 1-6

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for subjects with early ALS:

* Probable or definite ALS according to World Federation of Neurology diagnostic criteria4.
* Early stage ALS defined as presence of:

  1. Normal lower extremities muscle strength (≥ 4/5 in manual muscle strength or ≥ 80% in the computerized dynamometer quantitative muscle strength);
  2. ALSFRS score of ≥ than 30;
  3. FVC of ≥75% predicted;
  4. Ambulatory without the use of any assistive device.
* 18 - 75 years of age.
* Able to provide informed consent.

Inclusion Criteria for control subjects:

* Healthy 18 - 75 years of age without significant medical condition as defined by the investigator.
* Able to provide informed consent.
* Not having any of the exclusion criteria listed below.

Exclusion Criteria:

* Age < 18 or > 75 years.
* History of falls (2 or more in the last year), history of fainting, history of cerebrovascular accident (CVA) or myocardial infarction (MI), history of lower limb joint replacement.
* History of neuromuscular dysfunction "except diagnosis of ALS for individuals with ALS".
* Post-traumatic, septic, inflammatory, or neuropathic arthritis.
* Lower extremity injury/surgery that may effect balance.
* Vestibular pathology (i.e., inner ear problems, vertigo, meniere's).
* Peripheral neuropathy.
* Parkinson's Disease.
* Currently taking anti-convulsive medications (e.g., clonazepam, diazepam, lorazepam,phenytoin, zonegran, carbamazepine, depakote, gabapentin, lamotrigine, lamotrigine, oxcarbazepine, tiagabine, topiramate)
* Diabetes Mellitus.
* No history of neurological or medical condition that may interfere with balance as defined by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Amyotrophic Lateral Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
SOT equilibrium scores on conditions 1-6. | 9 monthes

SECONDARY OUTCOMES:
MSS on conditions 1-6 Weight Symmetry Score on conditions 1-6 DGI score TUG score POMA-B score | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sanjak, PhD, PT, MBA, Principal Investigator — Carolinas Healthcare Sysetm
Locations (1):
- Carolinas ALS Clinical Research Center, Charlotte, North Carolina, United States